CLINICAL TRIAL: NCT05169827
Title: How Cerebral Plasticity Shapes Symptom Progression in Parkinson's Disease: a Longitudinal Neuroimaging Study
Brief Title: Cerebral Contributions to Symptom Progression in PD
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL67597.091.18
Record Dates: First submitted 2021-03-30; First posted 2021-12-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: magnetic resonance imaging; motor assessment; symptom progression; action selection; compensation; basal ganglia
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PD-OFF: Patients with PD who have previously been included in the Personalized Parkinson Project return for fMRI measurements in an off-medicated state (12h withdrawal). N = 60.
  The PD-OFF group undergoes a single testing session.
- Healthy controls: Healthy individuals who are matched on age and sex with respect to the PD-OFF group. N = 60.
  The healthy group undergoes baseline and two year follow-up testing sessions.
- PD-ON: Patients with PD who are included in the Personalized Parkinson Project. N = 360.
  Available data will be used. There will be no further data collection in this group.

SUMMARY:
Motor symptom progression in early-stage Parkinson's disease varies substantially between individual patients. This progression correlates poorly with striatal dopamine depletion, which is largely complete four years post-diagnosis. Identification of alternative mechanisms, such as cortical compensatory processes, may enable more accurate predictions of individual motor progression.

DETAILED DESCRIPTION:
Striatal dopamine depletion leads to dysfunction in the cortico-striatal motor circuit and is an important contributor to motor symptoms in Parkinson's disease (PD). However, dopamine depletion in striatal motor regions is already severe at symptom onset and tends to correlate poorly with progressive worsening. This indicates that the severity of motor symptoms in PD may not be solely dependent on basal ganglia dysfunction. In PD, the deleterious effect of basal ganglia dysfunction on motor control may be partially counteracted by neuroplasticity and the compensatory recruitment of parieto-premotor areas of cortex that drive movement based on sensory cueing and goal-directed cognitive control. The efficacy of cortical compensation could therefore be a core determinant of motor impairment in PD.

This study utilizes longitudinal clinical and brain imaging data from early-stage PD patients included in the Personalized Parkinson Project (ClinicalTrials.gov Identifier: NCT03364894) to test whether motor symptom severity and progression can be predicted by action selection-related brain activity in parieto-premotor cortex, basal ganglia, or a combination of both.

Additional control analyses will be performed to investigate the effects of disease and medication on action selection-related brain activity. Action selection-related brain activity will be compared between PD patients and a cohort of healthy controls to assess the effect of disease (PD vs Healthy). Effects of medication (on vs. off) on action selection-related brain activity will be investigated through within-subject comparisons in subset of PD patients who underwent functional brain imaging in both on- and off-medicated states.

ELIGIBILITY:
Inclusion Criteria (patients):

* Subject is included in the Personalized Parkinson Project and has already participated in all baseline measurements (this means that inclusion and exclusion criteria of the Personalized Parkinson Project have already been fulfilled)
* Subject has completed the Informed Consent Form, as approved by the Ethics Committee

Exclusion Criteria (patients):

* Subject is not taking dopaminergic medication

Inclusion Criteria (healthy controls):

* Subject is at least 40 years old
* Subject can read and understand Dutch
* Subject has completed the Informed Consent Form, as approved by the Ethics Committee
* Subject is willing, competent, and able to comply with all aspects of the protocol, including follow-up schedule.

Exclusion Criteria (healthy controls):

* Subject has no co-morbidities that would negatively influence the interpretability of results from a comparison with PD patients (e.g. other neurodegenerative diseases or mental health disorders)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any person with, or without, Parkinson's disease who meets the inclusion criteria and does not meet the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Mid-term disease progression in terms of overall motor symptoms | Baseline and 2 years
  Change in Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III score, measured in off state. This scale assesses 18 motor symptoms (33 items) that are specific for Parkinson's disease. Item scores range from 0 to 4 and are summed, resulting in a total score ranging from 0 to 132, with higher scores representing worse outcomes.
Mid-term disease progression in terms of bradykinesia and rigidity | Baseline and 2 years
  Change in Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III score, measured in off state. This scale assesses 18 motor symptoms (33 items) that are specific for Parkinson's disease. Item scores range from 0 to 4. 17 items assessing bradykinesia and rigidity and are summed, resulting in a total score ranging from 0 to 68, with higher scores representing worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rick C Helmich, MD, PhD, Principal Investigator — Donders Centre for Cognitive Neuroimaging; Bastiaan R Bloem, MD, PhD, Principal Investigator — Radboud University Medical Center, Department of Neurology
Locations (1):
- Donders institute for brain, cognition and behaviour, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
See plan description for the Personalized Parkinson Project.
  In addition to these steps, we will make our statistical analysis plan and analytic code available to researchers that specifically focus on data related to the action selection task.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: TBA.
Access Criteria: Currently no list of criteria is available.

REFERENCES:
- [Background] Buhmann C, Binkofski F, Klein C, Buchel C, van Eimeren T, Erdmann C, Hedrich K, Kasten M, Hagenah J, Deuschl G, Pramstaller PP, Siebner HR. Motor reorganization in asymptomatic carriers of a single mutant Parkin allele: a human model for presymptomatic parkinsonism. Brain. 2005 Oct;128(Pt 10):2281-90. doi: 10.1093/brain/awh572. Epub 2005 Jun 9. PMID 15947065
- [Background] Helmich RC, de Lange FP, Bloem BR, Toni I. Cerebral compensation during motor imagery in Parkinson's disease. Neuropsychologia. 2007 Jun 11;45(10):2201-15. doi: 10.1016/j.neuropsychologia.2007.02.024. Epub 2007 Mar 7. PMID 17448507
- [Background] Herz DM, Eickhoff SB, Lokkegaard A, Siebner HR. Functional neuroimaging of motor control in Parkinson's disease: a meta-analysis. Hum Brain Mapp. 2014 Jul;35(7):3227-37. doi: 10.1002/hbm.22397. Epub 2013 Oct 5. PMID 24123553
- [Background] Herz DM, Meder D, Camilleri JA, Eickhoff SB, Siebner HR. Brain Motor Network Changes in Parkinson's Disease: Evidence from Meta-Analytic Modeling. Mov Disord. 2021 May;36(5):1180-1190. doi: 10.1002/mds.28468. Epub 2021 Jan 11. PMID 33427336
- [Background] Kordower JH, Olanow CW, Dodiya HB, Chu Y, Beach TG, Adler CH, Halliday GM, Bartus RT. Disease duration and the integrity of the nigrostriatal system in Parkinson's disease. Brain. 2013 Aug;136(Pt 8):2419-31. doi: 10.1093/brain/awt192. PMID 23884810
- [Background] Michely J, Volz LJ, Barbe MT, Hoffstaedter F, Viswanathan S, Timmermann L, Eickhoff SB, Fink GR, Grefkes C. Dopaminergic modulation of motor network dynamics in Parkinson's disease. Brain. 2015 Mar;138(Pt 3):664-78. doi: 10.1093/brain/awu381. Epub 2015 Jan 6. PMID 25567321
- [Background] van Nuenen BF, Helmich RC, Buenen N, van de Warrenburg BP, Bloem BR, Toni I. Compensatory activity in the extrastriate body area of Parkinson's disease patients. J Neurosci. 2012 Jul 11;32(28):9546-53. doi: 10.1523/JNEUROSCI.0335-12.2012. PMID 22787040
- [Background] van Nuenen BF, van Eimeren T, van der Vegt JP, Buhmann C, Klein C, Bloem BR, Siebner HR. Mapping preclinical compensation in Parkinson's disease: an imaging genomics approach. Mov Disord. 2009;24 Suppl 2:S703-10. doi: 10.1002/mds.22635. PMID 19877238
- [Background] Obeso JA, Rodriguez-Oroz MC, Rodriguez M, Lanciego JL, Artieda J, Gonzalo N, Olanow CW. Pathophysiology of the basal ganglia in Parkinson's disease. Trends Neurosci. 2000 Oct;23(10 Suppl):S8-19. doi: 10.1016/s1471-1931(00)00028-8. PMID 11052215
- [Background] Palop JJ, Chin J, Mucke L. A network dysfunction perspective on neurodegenerative diseases. Nature. 2006 Oct 19;443(7113):768-73. doi: 10.1038/nature05289. PMID 17051202
- [Background] Pirker W, Holler I, Gerschlager W, Asenbaum S, Zettinig G, Brucke T. Measuring the rate of progression of Parkinson's disease over a 5-year period with beta-CIT SPECT. Mov Disord. 2003 Nov;18(11):1266-72. doi: 10.1002/mds.10531. PMID 14639666
- [Background] Redgrave P, Rodriguez M, Smith Y, Rodriguez-Oroz MC, Lehericy S, Bergman H, Agid Y, DeLong MR, Obeso JA. Goal-directed and habitual control in the basal ganglia: implications for Parkinson's disease. Nat Rev Neurosci. 2010 Nov;11(11):760-72. doi: 10.1038/nrn2915. Epub 2010 Oct 14. PMID 20944662
- See also: Clinicaltrials.gov profile of the Personalized Parkinson Project — https://clinicaltrials.gov/ct2/show/NCT03364894?term=Personalized+Parkinson&draw=2&rank=1